CLINICAL TRIAL: NCT02925845
Title: Neuromuscular Electrostimulation Effect on the Maturation of Native Vascular Access (VA) Patients With Kidney Disease 5- Chronic Stages 5d Estimated by Doppler Ultrasound
Brief Title: Neuromuscular Electrostimulation in Radiocephalic Fistula
Acronym: NMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Terrassa (Other)
Responsible Party: Principal Investigator, Lucia Martínez Carnovale, Medical Doctor, Hospital de Terrassa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VES-COMPAVI-2014-01
Record Dates: First submitted 2016-09-29; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular electrostimulation (Experimental): Patients assigned to the group NMS, following the visit Day Hospital, in the first two hours of each HD session will perform a program of neuromuscular electrostimulation of the limb with the RC-AVF performed in the reference position of the flexors and extensors forearm at the tip intervened in each HD session on the stage previously established in the protocol (duration according to established program).
  Interventions: Device: Neuromuscular electrostimulation
- Isometric exercises (No Intervention): They will perform isometric exercises operated limb on an outpatient basis (repeated pressure rubber balls, heavy lifting 1-2 kg).

INTERVENTIONS:
Device: Neuromuscular electrostimulation — The device CompexTheta 400i provided with various developmental programs rehabilitation exercise with different phases, types and current is used. an adaptive program (heating, toning, muscular atrophy, strength-endurance) will be established for each patient during the study period. It shall apply at the level of the muscle bellies of the flexor and extensor muscles of the forearm dela upper extremity AV created. Electrodes are positioned at the anatomical reference positions. The intensity of the current will increase until a tolerable muscle contraction and painless by the patient.
  Arms: Neuromuscular electrostimulation

SUMMARY:
* Objective: To analyze the effect of neuromuscular electrostimulation in the maturation of radiocephalic arteriovenous fistula (RC-AVF) patients with chronic kidney disease (CKD) stage 5-5D
* Design: Clinical Trial with medical devices, 18-month, single-center, within the hospital setting.
* Disease or disorder study: vascular Access maturation.
* Population: Patients with CKD stage 5-5D at the research center.
* Project duration: 78 weeks
* Methodology:
* Patients with CKD stages 5-5D that has undergone a native AV in service stations to give their informed consent and meeting the inclusion criteria will be included.
* At baseline two study groups were established:

  * Group 1: neuromuscular electrostimulation
  * Group 2: isometric exercises

DETAILED DESCRIPTION:
* Objective: To analyze the effect of neuromuscular electrostimulation in the maturation of radiocephalic arteriovenous fistula (RC-AVF) patients with chronic kidney disease (CKD) stage 5-5D
* Design: Clinical Trial with medical devices, 18-month, single-center, within the hospital setting.
* Disease or disorder study: vascular Access maturation.
* Population: Patients with CKD stage 5-5D at the research center.
* Project duration: 78 weeks
* Methodology:
* Patients with CKD stages 5-5D that has undergone a native AV in service stations to give their informed consent and meeting the inclusion criteria will be included.
* At baseline two study groups were established:

  * Group 1: neuromuscular electrostimulation
  * Group 2: isometric exercises
* At baseline, patients included in the study the main demographic variables were collected, anthropometric, biochemical parameters, hemodynamic data, Eco Doppler of AV (ECO mapping) and prescribed medical treatment.
* Likewise, they will be made an assessment of their muscle strength by skinfold and upper limb static dynamometry in which was made the native AV.
* During the study period the following phases were established:

  • Phase 1 (4 weeks):
* The control group will receive the usual care on an outpatient AV.
* Patients assigned to group, will perform a program of AV electrostimulation in the affected upper extremity (according to program) after 7 days of completion of native AV.
* At the end of this phase both groups were conducted an ECO doppler (ECO4s) AV regulated by Vascular Surgery.

  • Phase 2 (8 weeks):
* The control group will receive the usual care on an outpatient AV.
* Patients assigned to group, will perform a program of AV electrostimulation in the affected upper extremity (according to program)
* At the end of this phase, both groups were conducted an ECO doppler (ECO8s) is regulated by the AV Vascular Surgery
* During all phases of the study, patients on hemodialysis follow their analytical controls programmed by Nephrology and receive medical treatment according to standard clinical practice.
* At the end of each phase of the study, all patients were performed an assessment of their muscle strength by centimetría, skinfold thickness and static dynamometry member in which AV has been made.
* Calendar: A provisional timetable is presented

  * Presentation of the CEIC study: September 2014
  * inclusion Period: 78 weeks
  * Follow-up period: 2 months
  * Close database: 1 month
  * Statistical analysis: 1 month
* Source of funding: Not available

ELIGIBILITY:
* Inclusion criteria:

  * Patients aged less than 18 years old
  * Patients with tracking CCEE Nephrology than 3 months
  * Patients with AV native AV upper limb without prior
  * Patients give their written informed consent
* Exclusion criteria:

  * prior cardiovascular event (acute myocardial infarction, unstable angina, stroke ....) in the last 3 months.
  * AV prior to HD in same upper extremity
  * Not have given informed written consent
  * Carrier cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Radiocephalic fístula flow ( millimeters/minuts) | 8 weeks ultrasonography parameter of maturation

SECONDARY OUTCOMES:
Complications related to radiocephalic fistula: thrombosis, haematoma, stenosis, early failure, reintervention | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lucía Inés Martínez Carnovale, MD, Principal Investigator — Hospital de Terrassa CST
Locations (1):
- Lucía Inés Martínez Carnovale, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brescia MJ, Cimino JE, Appell K, Hurwich BJ, Scribner BH. Chronic hemodialysis using venipuncture and a surgically created arteriovenous fistula. 1966. J Am Soc Nephrol. 1999 Jan;10(1):193-9. No abstract available. PMID 9890327
- [Background] Leaf DA, MacRae HS, Grant E, Kraut J. Isometric exercise increases the size of forearm veins in patients with chronic renal failure. Am J Med Sci. 2003 Mar;325(3):115-9. doi: 10.1097/00000441-200303000-00003. PMID 12640286
- [Background] Fontsere N, Mestres G, Yugueros X, Lopez T, Yuguero A, Bermudez P, Gomez F, Riambau V, Maduell F, Campistol JM. Effect of a postoperative exercise program on arteriovenous fistula maturation: A randomized controlled trial. Hemodial Int. 2016 Apr;20(2):306-14. doi: 10.1111/hdi.12376. Epub 2015 Oct 20. PMID 26486682